CLINICAL TRIAL: NCT00413231
Title: The Valiant Thoracic Stent Graft System. The Evaluation of the Clinical Performance of the Valiant Thoracic Stent Graft System in the Treatment of Descending Thoracic Aneurysms of Degenerative Etiology in Subjects Who Are Candidates for Endovascular Repair.
Brief Title: Valor II: The Valiant Thoracic Stent Graft System Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Investigational Plan #078
Record Dates: First submitted 2006-12-15; First posted 2006-12-19 (Estimated); Results first posted 2012-04-05 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Thoracic Aortic Aneurysm
Keywords: Thoracic Aneurysm; Endovascular Aortic Repair (EVAR); Endovascular Stent Graft; Endograft; Thoracic Aortic Aneurysm; Endovascular procedure; Descending Thoracic Aneurysm; Valiant Stent Graft System
MeSH Terms: conditions — Aortic Aneurysm, Thoracic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Valiant Thoracic Stent Graft System (Experimental): 160 subjects were enrolled into the study, including 157 subjects treated with the study device and three subjects classified as intent-to-treat who did not receive the study device.
  There were no other arms for this study.
  Interventions: Device: Valiant Thoracic Stent Graft System

INTERVENTIONS:
Device: Valiant Thoracic Stent Graft System — Surgical procedure in which a device is implanted inside the aorta, isolating the diseased area (aneurysm).
  Other Names: Valiant device; Valiant stent graft.

SUMMARY:
This study was designed to study safety and effectiveness of the Valiant Thoracic Stent Graft to treat thoracic aortic aneurysms.

DETAILED DESCRIPTION:
The aorta is a large blood vessel that carries blood away from the heart to the organs in the rest of the body. An aneurysm is a weakening in the artery wall that will become a bulge in the aorta. If left untreated, this bulge may continue to grow larger and may rupture (break open) with fatal consequences. In this research study we are investigating a device that can be placed in the aorta to exclude the weakened part of the artery wall and restore blood flow. Information will be collected on the performance of the device for 5 years.

ELIGIBILITY:
The following inclusion/exclusion criteria was obtained from the study protocol.

INCLUSION CRITERIA

To be eligible for enrollment, a subject must meet all of the following inclusion criteria:

1. Subject is between the age of 18 and 85.
2. Subject must be considered a candidate for elective surgical repair of the TAA (i.e., low-to-moderate risk [categories 0, 1, and 2] per the modified SVS/AAVS scoring system at the time of implant). See Appendix B: Modified SVS/AAVS Medical Co-Morbidity Grading System
3. If subject is female of childbearing potential, she must have a negative pregnancy test within 7 days before the implant procedure.
4. Subject has a DTA that is:

   1. A fusiform aneurysm with a maximum diameter of ≥ 5 cm OR is > 2 times the diameter of the non-aneurysmal thoracic aorta;

      AND/OR
   2. Saccular aneurysm (penetrating atherosclerotic ulcer)
5. Subject's anatomy must meet all of the following anatomical criteria:

   1. Subject's TAA must be ≥ 20 mm distal to the origin of the left common carotid artery and must be ≥ 20 mm proximal to the celiac artery;
   2. Proximal and distal non-aneurysmal neck diameter measurements must be between 20 mm and 42 mm;
   3. Proximal and distal non-aneurysmal neck must be ≥ 20 mm in length.
6. Thoracic aortic lesion is confirmed, at a minimum, by diagnostic contrast enhanced computerized tomography (CT) with optional 3-D reconstruction, and/or contrast enhanced Magnetic Resonance Angiogram obtained within four (4) months prior to the implant procedure.
7. Subject is able and willing to comply with the protocol and undergo follow-up requirements.
8. Subject or subject's legal representative understands and has signed an Informed Consent approved by the Sponsor and by the IRB for this study.
9. Subject has patent iliac or femoral arteries or can tolerate a vascular conduit that allows endovascular access to the aneurysmal site with the delivery system of the appropriate size device chosen for treatment.

EXCLUSION CRITERIA

To be eligible for enrollment, a subject cannot meet any of the following exclusion criteria:

1. Planned placement of the COVERED portion of the stent graft requires implant to occur in zones 0 or 1.
2. Subject has a thoracic aneurysm with a contained rupture.
3. Subject has a connective tissue disease (e.g., Marfan's syndrome, aortic medial degeneration).
4. Subject has a mycotic aneurysm or is suspected of having systemic infection.
5. Subject has received a previous stent or stent graft or previous surgical repair in the DTA.
6. Subject requires treatment of an infra-renal aneurysm at the time of implant.
7. Subject has a history of bleeding diathesis, coagulopathy, or refuses blood transfusion.
8. Subject has had or plans to have a major surgical procedure within 30 days before or after the Valiant Stent Graft procedure. This does not include planned procedures that are needed for the safe and effective placement of the stent graft (i.e., carotid/subclavian transposition, carotid/subclavian bypass procedure).
9. Subject has had an MI or cerebral vascular accident (CVA) within 3 months.
10. Subject is currently participating in an investigational drug or device clinical trial.
11. Subject has a known allergy or intolerance to the device components.
12. Subject has a known hypersensitivity or contraindication to anticoagulants or contrast media, which is not amenable to pre-treatment.
13. Subject has significant and/or circumferential aortic mural thrombus at either the proximal or distal attachment sites that would compromise fixation and seal of the device.
14. Subject has other medical, social, or psychological problems that, in the opinion of the investigator, preclude him or her from receiving this treatment and the procedures and evaluations pre- and post-treatment, or a limited life expectancy of less than 1 year.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2006-12; Primary Completion 2010-08 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Fairman, MD, Principal Investigator — University of Pennsylvania
Locations (26):
- United States (26):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Southern California - Healthcare Consultation Center, Los Angeles, California
  - Los Angeles Biomedical Research Institute @ Harbor-UCLA Medical Center, Torrance, California
  - Hartford Hospital, Hartford, Connecticut
  - University of Florida, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - Union Memorial, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - Minneapolis Vascular Physicians, Plymouth, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Advance Vascular Associates (Morristown Memorial Hospital), Morristown, New Jersey
  - Albany Medical Center, Albany, New York
  - New York University Medical Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Shadyside Hospital - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - St. Luke's Episcopal Hospital - Houston, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia

REFERENCES:
- [Derived] Conrad MF, Tuchek J, Freezor R, Bavaria J, White R, Fairman R. Results of the VALOR II trial of the Medtronic Valiant Thoracic Stent Graft. J Vasc Surg. 2017 Aug;66(2):335-342. doi: 10.1016/j.jvs.2016.12.136. Epub 2017 Mar 30. PMID 28366302

RESULTS

PARTICIPANT FLOW:
Groups:
- Valiant Thoracic Stent Graft System: Subjects treated or intended to treat with the test device (Valiant Thoracic Stent Graft System).
Period: 0 to 30-day Post Treatment
Arm/Group | Valiant Thoracic Stent Graft System
Started | 160
Completed | 152
Not Completed | 8
Not completed — Death | 5
Not completed — Intend to treat, but not implanted | 3
Period: 30-day to 365-day Post Treatment
Arm/Group | Valiant Thoracic Stent Graft System
Started | 152
Completed | 139
Not Completed | 13
Not completed — Death | 13
Period: 365-day to 60-month Post Treatment
Arm/Group | Valiant Thoracic Stent Graft System
Started | 139
Completed | 93
Not Completed | 46
Not completed — Death | 36
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 4
Not completed — Exited after surgical conversion | 1

BASELINE CHARACTERISTICS:
Arm/Group | Valiant Thoracic Stent Graft System
Number analyzed (Participants) | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.2 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 95
Region of Enrollment [Number; unit: participants]
  United States | 160

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants That Did NOT Experience Aneurysm-Related Mortality (Post-market Primary Endpoint)
Description: Evaluation of the ARM-free rate in subjects implanted with the Valiant Thoracic Stent Graft five years post-implantation by comparing it to a pre-defined performance goal (PG) based on an analysis of ARM-free rates from TEVAR data and on results from the VALOR (Talent Thoracic Endoluminal Stent Graft, IDE G980116) clinical study.
Time Frame: 0 through 1825 days post treatment
Population: Subjects treated or intended to treat with the test device
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Valiant Thoracic Stent Graft System
Number analyzed (Participants) | 160
Percentage of participants | 94.8 [90.9 to 97.1]

2. Secondary Outcome: Percentage of Subjects That Experienced Successful Deployment and Delivery of the Stent Graft at Implant
Description: Percentage of subjects that experienced successful deployment and delivery of the stent graft at implant. Successful deployment and delivery of the stent graft is used to measure effectiveness.
Time Frame: At implant
Population: Subjects treated or intended to treat with the test device
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Valiant Thoracic Stent Graft System: 160 subjects were enrolled into the study, including 157 subjects treated with the study device and three subjects classified as intent-to-treat who did not receive the study device.
  There were no other arms for this study.
  Valiant Thoracic Stent Graft System: Surgical procedure in which a device is implanted inside the aorta, isolating the diseased area (aneurysm).
Arm/Group | Valiant Thoracic Stent Graft System
Number analyzed (Participants) | 160
Percentage of participants | 96.3 [92 to 98.6]

3. Secondary Outcome: Percentage of Participants That Experienced Perioperative Mortality
Description: Percentage of subjects that experienced perioperative mortality. Perioperative morality is defined as all-cause mortality within 30 days after index procedure.
Time Frame: Within 30 days post treatment
Population: Subjects treated or intended to treat with the test device
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Valiant Thoracic Stent Graft System
Number analyzed (Participants) | 160
Percentage of participants | 3.1 [1 to 7.1]

4. Secondary Outcome: Percentage of Participants That Experienced Paraplegia
Description: Percentage of subjects that experienced paraplegia within 30 days post treatment
Time Frame: Within 30 days post treatment
Population: Subjects treated or intended to treat with the test device
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Valiant Thoracic Stent Graft System
Number analyzed (Participants) | 160
Percentage of participants | 0.6 [0 to 3.4]

5. Primary Outcome: Percentage of Participants With Successful Aneurysm Treatment (Primary Effectiveness Endpoint)
Description: Percentage of subjects with absence of both: a) aneurysm growth of more than 5 mm at the 12-month visit relative to the 1-month visit; and b) secondary procedure due to type I or III endoleak performed or recommended at or before the 12-month visit. Success means a subject experienced neither a nor b.
  Type I: endoleak in continuity with the proximal anchoring site(proximal endoleak) or the distal anchoring site(distal endoleak)of the device.
  Type III: endoleak is present in the mid-graft region due to defect of fabric or between the segments of the modular graft (junctional endoleak).
Time Frame: At 12-month post procedure
Population: Subjects treated or intended to treat with the test device
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Valiant Thoracic Stent Graft System
Number analyzed (Participants) | 160
Percentage of Participants | 97.4 [93.4 to 100]

6. Primary Outcome: Percentage of Participants Who Died (Primary Safety Endpoint: All-Cause Mortality) > >
Description: The percentage of participants who died within 12-months of the initial procedure, whether or not the cause of death was related to the study device, procedure, or condition treated.
  >
  > Note: All-cause mortality endpoint is not directly related to successful aneurysm treatment, which pertains to the absence of aneurysm growth and secondary procedure due to Type I and III endoleaks.
Time Frame: Within 12-months post treatment
Population: Subjects treated or intended to treat with the test device
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Valiant Thoracic Stent Graft System
Number analyzed (Participants) | 160
Percentage of Participants | 12.6 [7.3 to 17.9]

7. Secondary Outcome: Percentage of Participants That Experienced Paraparesis
Description: Percentage of subjects that experienced paraparesis within 30 days post treatment
Time Frame: Within 30 days post treatment
Population: Subjects treated or intended to treat with the test device
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Valiant Thoracic Stent Graft System
Number analyzed (Participants) | 160
Percentage of participants | 1.9 [0.4 to 5.4]

8. Secondary Outcome: Percentage of Participants That Experienced Secondary Procedures Due to Endoleak After Discharge
Description: Percentage of subjects that experienced secondary procedures due to endoleak after discharge within 30 days post treatment
Time Frame: Within 30 days post treatment
Population: Subjects treated or intended to treat with the test device
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Valiant Thoracic Stent Graft System
Number analyzed (Participants) | 160
Percentage of participants | 0.6 [0 to 2.5]

9. Secondary Outcome: Percentage of Participants That Experienced One or More Major Adverse Events
Description: Percentage of subjects that experienced one or more major adverse events within 30 days post treatment, regardless of relatedness to study device
Time Frame: Within 30 days post treatment
Population: Subjects treated or intended to treat with the test device
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Valiant Thoracic Stent Graft System
Number analyzed (Participants) | 160
Percentage of participants | 38.1 [30.6 to 46.1]

10. Secondary Outcome: Percentage of Participants That Experienced Aneurysm-related Mortality
Description: Percentage of subjects that experienced aneurysm-related mortality within 12 months post treatment
Time Frame: Within 12 months post treatment
Population: Subjects treated or intended to treat with the test device, excluding subjects exited before 12 months and implant failures
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Valiant Thoracic Stent Graft System
Number analyzed (Participants) | 151
Percentage of participants | 3.3 [1.1 to 7.6]

11. Secondary Outcome: Percentage of Participants That Experience Aneurysm Rupture
Description: Percentage of subjects that experience aneurysm rupture within 12 months post treatment
Time Frame: Within 12 months post treatment
Population: Subjects treated or intended to treat with the test device excluding subjects that exited before 12 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Valiant Thoracic Stent Graft System
Number analyzed (Participants) | 154
Percentage of participants | 0 [0 to 2.4]

12. Secondary Outcome: Percentage of Participants That Experienced Conversion to Open Surgical Repair
Description: Percentage of subjects that experienced conversion to open surgical repair within 12 months post treatment
Time Frame: Within 12 months post treatment
Population: Subjects treated or intended to treat with the test device excluding subjects exited before 12 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Valiant Thoracic Stent Graft System
Number analyzed (Participants) | 154
Percentage of participants | 0 [0 to 2.4]

13. Secondary Outcome: Percentage of Participants That Experienced Endoleak(s)
Description: Percentage of subjects that experienced endoleak(s) of any type at 12 months
Time Frame: At 12 months
Population: Subjects treated or intended to treat with the test device excluding subjects that did not have proper imaging to identify endoleaks
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Valiant Thoracic Stent Graft System
Number analyzed (Participants) | 100
Percentage of participants | 13 [7.1 to 21.2]

14. Secondary Outcome: Percentage of Participants That Experienced Secondary Endovascular Procedures Due to Endoleak
Description: Percentage of subjects that experienced secondary endovascular procedures due to endoleak between 30 days and 12 months
Time Frame: Between 30 days and 12 months
Population: Subjects treated or intended to treat with the test device excluding censored subjects (those with no data within the time frame)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Valiant Thoracic Stent Graft System
Number analyzed (Participants) | 143
Percentage of participants | 0 [0 to 2.5]

15. Secondary Outcome: Percentage of Participants That Experienced Stent Graft Migration
Description: Percentage of subjects that experienced stent graft migration within 12 months post treatment, as reported by the CEC. Of note, all migrations resulted from anatomical accommodation of the stent graft. All migrations were at the distal end of the stent graft, moving proximally. No endoleaks were associated to these migrations.
Time Frame: Within 12 months post treatment
Population: Subjects treated or intended to treat with the test device, excluding subjects that did not have proper imaging
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Valiant Thoracic Stent Graft System
Number analyzed (Participants) | 105
Percentage of participants | 2.9 [0.6 to 8.1]

16. Secondary Outcome: Percentage of Participants That Experience Loss of Stent Graft Patency
Description: Percentage of subjects that experience loss of stent graft patency within 12 months post treatment
Time Frame: Within 12 months post treatment
Population: Subjects treated or intended to treat with the test device, excluding subjects that did not have proper imaging
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Valiant Thoracic Stent Graft System
Number analyzed (Participants) | 100
Percentage of participants | 0 [0 to 3.6]

17. Secondary Outcome: Percentage of Participants That Experienced One or More Major Adverse Events
Description: Percentage of subjects that experienced one or more Major Adverse Events within 12 months post treatment
Time Frame: Within 12 months post treatment
Population: Subjects treated or intended to treat with the test device, excluded subjects that exited before 12 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Valiant Thoracic Stent Graft System
Number analyzed (Participants) | 154
Percentage of participants | 48.7 [40.6 to 56.9]

18. Secondary Outcome: Percentage of Participants That Died (All-cause Mortality)
Description: Percentage of subjects that died (all-cause mortality) five years post implant, regardless whether or not the cause of death was related to procedure, device, or condition treated
Time Frame: 0 through 1825 days post treatment
Population: Subjects treated or intended to treat with the test device
Measure: Number; unit: Percentage of participants
Arm/Group | Valiant Thoracic Stent Graft System
Number analyzed (Participants) | 160
Percentage of participants | 33.8

19. Secondary Outcome: Percentage of Participants That Experienced Aneurysm-related Mortality
Description: Percentage of subjects that experienced aneurysm-related within five years post implant
Time Frame: 0 through 1825 days post treatment
Population: Subjects treated or intended to treat with the test device
Measure: Number; unit: Percentage of participants
Arm/Group | Valiant Thoracic Stent Graft System
Number analyzed (Participants) | 160
Percentage of participants | 5

20. Secondary Outcome: Percentage of Participants That Experienced Aneurysm Ruptures
Description: Percentage of subjects that experienced aneurysm ruptures within five years post implant
Time Frame: 0 through 1825 days post treatment
Population: Subjects treated or intended to treat with the test device
Measure: Number; unit: Percentage of participants
Arm/Group | Valiant Thoracic Stent Graft System
Number analyzed (Participants) | 160
Percentage of participants | 1.3

21. Secondary Outcome: Percentage of Participants That Experienced Conversions to Open Surgical Repair
Description: Percentage of subjects that experienced conversions to open surgical repair within five years post implant
Time Frame: 0 through 1825 days post treatment
Population: Subjects treated or intended to treat with the test device
Measure: Number; unit: Percentage of participants
Arm/Group | Valiant Thoracic Stent Graft System
Number analyzed (Participants) | 160
Percentage of participants | 0.6

22. Secondary Outcome: Percentage of Participants That Experienced Type I Endoleaks
Description: Percentage of subjects that experienced type I endoleaks within five years post implant
Time Frame: 0 through 1825 days post treatment
Population: Subjects treated or intended to treat with the test device
Measure: Number; unit: Percentage of participants
Arm/Group | Valiant Thoracic Stent Graft System
Number analyzed (Participants) | 160
Percentage of participants | 8.1

23. Secondary Outcome: Percentage of Participants That Experienced Type III Endoleaks
Description: Percentage of subjects that experienced type III endoleaks within five years post implant
Time Frame: 0 through 1825 days post treatment
Population: Subjects treated or intended to treat with the test device
Measure: Number; unit: Percentage of participants
Arm/Group | Valiant Thoracic Stent Graft System
Number analyzed (Participants) | 160
Percentage of participants | 0.6

24. Secondary Outcome: Percentage of Participants That Experienced Type IV Endoleaks
Description: Percentage of subjects that experienced type IV endoleaks within five years post implant
Time Frame: 0 through 1825 days post treatment
Population: Subjects treated or intended to treat with the test device
Measure: Number; unit: Percentage of participants
Arm/Group | Valiant Thoracic Stent Graft System
Number analyzed (Participants) | 160
Percentage of participants | 1.3

25. Secondary Outcome: Percentage of Participants That Experienced Secondary Endovascular Procedures
Description: Percentage of subjects that experienced secondary endovascular procedures within five years post implant
Time Frame: 0 through 1825 days post treatment
Population: Subjects treated or intended to treat with the test device
Measure: Number; unit: Percentage of participants
Arm/Group | Valiant Thoracic Stent Graft System
Number analyzed (Participants) | 160
Percentage of participants | 6.9

26. Secondary Outcome: Percentage of Participants That Experienced Stent Graft Migrations (Site Reported)
Description: Percentage of subjects that experienced stent graft migrations within five years post implant, as reported by the clinical sites
Time Frame: 0 through 1825 days post treatment
Population: Subjects treated or intended to treat with the test device
Measure: Number; unit: Percentage of participants
Arm/Group | Valiant Thoracic Stent Graft System
Number analyzed (Participants) | 160
Percentage of participants | 0

27. Secondary Outcome: Percentage of Participants That Experienced Loss of Stent Graft Patency
Description: Percentage of subjects that experienced loss of stent graft patency within five years post implant
Time Frame: 0 through 1825 days post treatment
Population: Subjects treated or intended to treat with the test device
Measure: Number; unit: Percentage of participants
Arm/Group | Valiant Thoracic Stent Graft System
Number analyzed (Participants) | 160
Percentage of participants | 0

ADVERSE EVENTS:
Time Frame: 60 months
Arm/Group | Valiant Thoracic Stent Graft System
Serious Adverse Events (participants affected / at risk) | 135/160
Other Adverse Events (participants affected / at risk) | 160/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valiant Thoracic Stent Graft System (N=160)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3)
Abdominal hernia (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Anaemia (Blood and lymphatic system disorders) | 6 (7)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 7 (7)
Angina unstable (Cardiac disorders) | 3 (4)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Aortic aneurysm (Vascular disorders) | 22 (26) — Includes non-treated aneurysm, such as abdominal aneurysms, and aneurysm expansion of treated aneurysms
Aortic aneurysm rupture (Vascular disorders) | 2 (2)
Aortic dissection (Vascular disorders) | 5 (5)
Aortic rupture (Injury, poisoning and procedural complications) | 2 (2)
Aortic valve stenosis (Cardiac disorders) | 1 (1)
Arterial injury (Injury, poisoning and procedural complications) | 8 (8)
Arterial occlusive disease (Vascular disorders) | 3 (3)
Arteriosclerosis (Vascular disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Asbestosis (Injury, poisoning and procedural complications) | 1 (1)
Asthenia (General disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 8 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Bladder catheter replacement (Surgical and medical procedures) | 1 (1)
Blood lactic acid increased (Investigations) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 14 (16)
Cardio-respiratory arrest (Cardiac disorders) | 3 (3)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 6 (7)
Chest pain (General disorders) | 10 (16)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Clostridial infection (Infections and infestations) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colostomy closure (Surgical and medical procedures) | 2 (2)
Complication of device insertion (General disorders) | 1 (1)
Convulsion (Nervous system disorders) | 2 (2)
Coronary angioplasty (Surgical and medical procedures) | 1 (1)
Coronary artery disease (Cardiac disorders) | 3 (3)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Death (General disorders) | 1 (1) — Unknown cause of death. Overall in the study, there were 54 deaths (46 not related to the TAA; 8 related to the TAA). However, this death could not be classified any further, as site was unable to obtain any information associated to it.
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Device deployment issue (General disorders) | 2 (2)
Device related infection (Infections and infestations) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (3)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Encephalopathy (Nervous system disorders) | 1 (1)
Endocardial fibroelastosis (Cardiac disorders) | 1 (1)
Eyeball rupture (Injury, poisoning and procedural complications) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Femoral arterial stenosis (Vascular disorders) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (2)
Gangrene (Infections and infestations) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 12 (14)
Generalised oedema (General disorders) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin abscess (Infections and infestations) | 1 (1)
Haematoma (Vascular disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Haemorrhage intracranial (Nervous system disorders) | 4 (4)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Hernia repair (Surgical and medical procedures) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 3 (3)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypertensive emergency (Cardiac disorders) | 1 (1)
Hypotension (Vascular disorders) | 4 (5)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2)
Impaired healing (General disorders) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 2 (2)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Lymphocele (Vascular disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 3 (3)
Medical device complication (General disorders) | 1 (1) — Right prosthetic knee infection
Mental status changes (Psychiatric disorders) | 5 (5) — E.g., Confusion, aphasia, and disorientation
Metabolic acidosis (Metabolism and nutrition disorders) | 3 (3)
Multi-organ failure (General disorders) | 2 (2)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Myocardial infarction (Cardiac disorders) | 12 (14)
Nausea (Gastrointestinal disorders) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 4 (4)
Non-small cell lung cancer stage IIIB (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Open wound (Injury, poisoning and procedural complications) | 1 (1)
Operative haemorrhage (Injury, poisoning and procedural complications) | 6 (6)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Panic disorder (Psychiatric disorders) | 1 (1)
Paraparesis (Nervous system disorders) | 1 (1)
Paraplegia (Nervous system disorders) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 1 (1)
Peripheral artery dissection (Vascular disorders) | 1 (1)
Peripheral embolism (Vascular disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (9)
Pneumonia (Infections and infestations) | 12 (15)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Pneumonia herpes viral (Infections and infestations) | 1 (1)
Poor peripheral circulation (Vascular disorders) | 1 (1)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 3 (3)
Presyncope (Nervous system disorders) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1)
Pulmonary embolism (Reproductive system and breast disorders) | 5 (5)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 4 (5)
Renal failure acute (Renal and urinary disorders) | 7 (7)
Renal failure chronic (Renal and urinary disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 16 (19)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Sepsis (Infections and infestations) | 9 (11)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal cord ischaemia (Nervous system disorders) | 2 (2)
Splenic embolism (Vascular disorders) | 1 (1)
Stent-graft endoleak (General disorders) | 13 (17) — TAA endoleaks: Type I, 9 events; Type II, 3; Type V/Unknown, 3. AAA endoleaks: 2 events
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Systemic candida (Infections and infestations) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 5 (5)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (3)
Urinary tract infection pseudomonal (Infections and infestations) | 1 (2)
Varices oesophageal (Gastrointestinal disorders) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 1 (1)
Ventricular tachyarrhythmia (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Vessel puncture site haematoma (General disorders) | 4 (4)
Vocal cord paralysis (Nervous system disorders) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 2 (2)
arteriovenous fistula (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valiant Thoracic Stent Graft System (N=160)
Abdominal Pain (Gastrointestinal disorders) | 8 (10)
Aortic aneurysm (Vascular disorders) | 14 (17) — Includes non-treated aneurysm, such as abdominal aneurysms, and aneurysm expansion of treated aneurysms
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Atrial fibrillation (Cardiac disorders) | 22 (24)
Back Pain (Musculoskeletal and connective tissue disorders) | 32 (35)
Chest pain (General disorders) | 21 (28)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Haematocrit decreased (Investigations) | 9 (9)
Headache (Nervous system disorders) | 8 (8)
Hypertension (Vascular disorders) | 15 (15)
Mental status changes (Psychiatric disorders) | 19 (21) — E.g. Confusion, worsening memory, and anxiety
Nausea (Gastrointestinal disorders) | 11 (11)
Oedema peripheral (General disorders) | 9 (9)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 17 (17)
Pneumonia (Infections and infestations) | 8 (8)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 8 (8)
Pyrexia (General disorders) | 17 (17)
Renal failure (Renal and urinary disorders) | 9 (9)
Stent-graft endoleak (General disorders) | 32 (37) — TAA endoleaks: Type I, 6 events; Type II, 20; Type III, 1; Type IV, 2; Type V/Unknown, 5. AAA endoleaks: 3 events.
Urinary tract infection (Infections and infestations) | 13 (16)
Vessel puncture site haematoma (General disorders) | 10 (10)

LIMITATIONS AND CAVEATS:
Adverse Events and Serious Adverse Events listed in ClinicalTrials.gov were re-coded, using MedDRA 13.1. To do so, events were reclassified. As a result, data in listings may not match those in Clinical Update reports, SSEDs, or Instructions for Use.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator (PI) and institution agree not to publish the results of the study until after the earliest of the following: a)conclusion of the study, b)the early termination of the study, c)at discretion and approval of the sponsor, or d)after sponsor confirms there will be no multicenter study publication, whichever occurs first. PI and institution further agree to submit to sponsor copies of any proposed publication or public presentation at least sixty days before dissemination.